CLINICAL TRIAL: NCT03752203
Title: Sodium Fluorescein-Guided Resection of Pediatric Neurosurgical Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study cancelled by PI.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-0242.cc
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Neurosurgical Tumors
Keywords: Sodium Fluorescein; Surgical Microscope; Central Nervous System; Tumors
MeSH Terms: conditions — Neoplasms | interventions — Fluorescein

STUDY DESIGN:
Intervention Model Description: The primary neurosurgeons who will perform the resections will be investigators on the study and will identify eligible patients from the established practice. At the time surgical intervention is recommended, the doctors will inform patients and parents/guardians of the existence of the study. Only those subjects with a clinical relationship to the study investigators will be recruited.
Masking Description: Since patients are being recruited from the investigators' practices, and there is only one form of treatment, masking will not be utilized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Sodium-Fluorescein Resection (Experimental): This study will employ the use of sodium fluorescein and an FDA approved operative microscope equipped with excitation and barrier filters for monitoring with sufficient fluorescent enhancement and contrast.
  Interventions: Drug: Sodium Fluorescein; Device: Microscopic Resection

INTERVENTIONS:
Drug: Sodium Fluorescein — Patients enrolled in this study will receive 3 mg/kg sodium fluorescein following induction of anesthesia by administration into a peripheral venous line over 10 seconds
Device: Microscopic Resection — Resection will proceed with the use of a surgical microscope equipped with excitation and barrier filters for monitoring with sufficient fluorescent enhancement and contrast.

SUMMARY:
Sodium fluorescein, which has been shown to be useful for intraoperative guidance regarding the resection of adult neurosurgical tumors, can aid the resection of pediatric neurosurgical tumors.

DETAILED DESCRIPTION:
This study will be a prospective non-randomized cohort study with patients presenting to Children's Hospital Colorado for resection of a central nervous system tumor. This study will employ the use of sodium fluorescein and an FDA approved operative microscope equipped with excitation and barrier filters for monitoring with sufficient fluorescent enhancement and contrast. Fluorescein sodium is a small organic salt that accumulates in areas of diminished blood-brain barrier integrity and allows for determination of the margins between tumor and normal brain function.

ELIGIBILITY:
Inclusion Criteria:

* Age 31 days through 21 years on date of surgery
* Undergoing resection of a central nervous system tumor at Children's Hospital Colorado
* Parent/legal guardian (or adult subject) willing and able to complete the informed consent process

Exclusion Criteria:

* Tumor in functionally eloquent cortex that precludes maximal surgical resection
* Severe renal dysfunction
* Preoperative serum creatinine level > than normal range and GFR < 30.
* Severe liver dysfunction
* History of asthma or pulmonary spasm
* Known allergy to sodium fluorescein or any other contrast dye
* Previous administration of sodium fluorescein within the last 72 hours
* Pregnant or nursing mother
* Other unspecified reasons that, in the opinion of the investigator, make the subject unsuitable for enrollment.

Ages: 31 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Hankinson, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium-Fluorescein Resection
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sodium-Fluorescein Resection
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent of Tumor Resected: Intracranial Lesions
Description: For all patients, pre-operative imaging and post-operative imaging will be used to analyze the extent of resection of the tumors. In intracranial lesions, the use of volumetric imaging tools will be used to calculate the extent of tumor resection.
Time Frame: Pre-op assessment to outpatient follow up, up to 6 weeks
Population: Data not collected or analyzed and therefore cannot be reported . Study was terminated due to lack of patients and funding. The Outcome Measure Data Table is not able to be completed due to lack of data.
Arm/Group | Sodium-Fluorescein Resection
Number analyzed (Participants) | 0

2. Primary Outcome: Percent of Tumor Resected: Spinal Lesions
Description: For all patients, pre-operative imaging and post-operative imaging will be used to analyze the extent of resection of the tumors. In spinal lesions, manual measurement will be used to determine the extent of resection.
Time Frame: Pre-op assessment to outpatient follow up, up to 6 weeks
Population: Data not collected.
Arm/Group | Sodium-Fluorescein Resection
Number analyzed (Participants) | 0

3. Post Hoc Outcome: No Outcome Measures Were Completed Due to Data Not Collected Due to Lack of Patients and Funding.
Description: No Outcome Measures were completed due to data not collected due to lack of patients and funding.
Time Frame: No Outcome Measures were completed due to data not collected due to lack of patients and funding.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Sodium-Fluorescein Resection
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Study was discontinued due to lack of funding and patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03752203/Prot_SAP_ICF_000.pdf